CLINICAL TRIAL: NCT00194103
Title: Effectiveness of Extended Telephone Monitoring
Acronym: ETM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Dr. James R McKay, PhD, University of Pennsylvania
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 708753; R01AA014850 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — Counseling

ARMS (3):
- TAU (No Intervention)
- Telephone Monitoring (Active Comparator)
  Interventions: Behavioral: Telephone Monitoring and Feedback
- Telephone Monitoring and Counseling (Experimental)
  Interventions: Behavioral: Telephone Monitoring and Counseling

INTERVENTIONS:
Behavioral: Telephone Monitoring and Feedback — In addition to attending IOP, participants receive phone contact from our counselors but only to receive a monitoring assessment. There is no feedback or counseling from study staff in this condition.
  Arms: Telephone Monitoring
Behavioral: Telephone Monitoring and Counseling — In addition to attending IOP, participants have phone contact with study counselors, which includes monitoring, feedback, and counseling.
  Arms: Telephone Monitoring and Counseling

SUMMARY:
The purpose of this study is to determine the effectiveness of extended telephone monitoring for alcohol-dependent patients receiving intensive outpatient treatment. It is hypothesized that telephone monitoring will produce better alcohol use outcomes relative to treatment as usual. It is also hypothesized that adaptive telephone monitoring plus brief counseling will produce better alcohol use outcomes over time relative to telephone monitoring plus feedback only.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in Intensive Outpatient substance abuse treatment for at least 2 and no more than 4 weeks at study entry
* qualify for a current DSM-IV diagnosis of alcohol dependence (during the month prior to entrance into the IOP or detoxification program prior to IOP);
* willingness to participate in research and be randomized;
* 4th grade reading level (as determined by the Slosson Oral Reading Test; Slosson, 1963);
* able to provide the names of several informants who will know his/her whereabouts during the follow-up period

Exclusion Criteria:

* acute medical or psychiatric problems that preclude outpatient treatment (e.g., in a psychotic episode and not stabilized on medication);
* IV heroin use during the past year;
* anticipated involvement in other forms of intensive treatment (e.g., inpatient) during the 6-month period after enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2004-05; Primary Completion 2009-08 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
TimeLineFollowBack | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: James McKay, Ph. D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States